CLINICAL TRIAL: NCT00309998
Title: Vinorelbine Plus Bevacizumab as First Line Therapy in Patients ≥ 70 Years of Age With Stage IIIB/IV Non-Squamous, Non-Small Cell Lung Cancer
Brief Title: Vinorelbine and Bevacizumab in Treating Older Patients With Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000465498; URCC-U1505; GENENTECH-AVF3328S
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; large cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Bevacizumab; Vinorelbine

INTERVENTIONS:
Biological: bevacizumab
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as vinorelbine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving vinorelbine together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving vinorelbine together with bevacizumab works in treating older patients with stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the median time to disease progression in older patients with non-squamous stage IIIB or stage IV non-small cell lung cancer (NSCLC) treated with vinorelbine ditartate and bevacizumab.

Secondary

* Estimate the response rate in patients treated with this regimen.
* Estimate the median survival in patients treated with this regimen.
* Evaluate the safety of the combination of vinorelbine ditartate and bevacizumab in older patients.

OUTLINE: This is an open-label study.

Patients receive vinorelbine ditartate IV over 6 to 10 minutes on days 1 and 8 and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days in the absence of unacceptable toxicity or disease progression.

After completion of study therapy, patients are followed periodically.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-squamous, non-small cell lung cancer (NSCLC)

  * Stage IIIB (any T, N3, M0 OR T4, any N, M0, OR pleural effusion) OR stage IV (any T, any N, M1) disease
  * Mixed tumors will be categorized by the predominant cell type unless small cell elements are present, in which case the patient is ineligible
* Measurable or evaluable disease
* No lung carcinoma of squamous cell histology or any histology in close proximity to a major vessel or cavitation
* No known brain metastases, even if treated

PATIENT CHARACTERISTICS:

* No other malignancies within the past 5 years except nonmelanoma skin cancer
* ECOG performance status 0-1
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 mg/dL
* Transaminases ≤ 5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN
* Urine protein:creatinine ratio < 1
* INR ≤ 1.5
* PTT normal
* No prior ileus or neuropathy compromising use of vinorelbine ditartate
* Patients with a history of hypertension must be well controlled (blood pressure < 150/100 mm Hg) on a stable regimen of antihypertensive therapy
* None of the following conditions:

  * Unstable angina
  * New York Heart Association grade II-IV congestive heart failure
  * Myocardial infarction within the past 6 months
  * Stroke within the past 6 months
  * Evidence of bleeding diathesis or coagulopathy
  * Clinically significant peripheral vascular disease
  * Serious, nonhealing wound, ulcer, or bone fracture
  * History of hemoptysis (bright red blood ≥ ½ teaspoon)
* No significant traumatic injury within the past 4 weeks
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for NSCLC
* More than 4 weeks since prior and no concurrent participation in another experimental drug study
* More than 4 weeks since prior immunotherapy, hormonal therapy, or radiotherapy and recovered
* More than 28 days since prior major surgical procedure or open biopsy

  * No anticipation of need for major surgery during course of trial
* More than 7 days since prior minor surgical procedures (e.g., fine-needle aspiration or core biopsy)
* No concurrent full-dose anticoagulation therapy for thromboembolic disease, aspirin (> 325 mg/day), or nonsteroidal anti-inflammatory drugs

Ages: 70 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-09; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Median time to disease progression by imaging study every 6 weeks

SECONDARY OUTCOMES:
Response rate by imaging study every 6 weeks
Median survival
Safety as measured by toxicity (e.g thromboembolism, bleeding, or bowel perforation) every three weeks or as required

CONTACTS AND LOCATIONS:
Overall Officials: Deepak M. Sahasrabudhe, MD, Study Chair — James P. Wilmot Cancer Center
Locations (1):
- James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York, United States